CLINICAL TRIAL: NCT01755507
Title: Double-blind,Randomized, Placebo-controlled, Phase II Dose-finding Study Comparing Different Doses of Norursodeoxycholic Acid Capsules With Placebo in the Treatment of Primary Sclerosing Cholangitis
Brief Title: Norursodeoxycholic Acid in the Treatment of Primary Sclerosing Cholangitis
Acronym: NUC-3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NUC-3/PSC
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Primary Sclerosing Cholangitis
Keywords: PSC
MeSH Terms: conditions — Cholangitis, Sclerosing

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- B (Experimental): norUDCA
  Interventions: Drug: norUDCA
- C (Experimental): norUDCA
  Interventions: Drug: norUDCA
- placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- A (Experimental): norUDCA
  Interventions: Drug: norUDCA

INTERVENTIONS:
Drug: norUDCA — Comparison of different dosages of norUDCA acid administered orally.
  Arms: A; B; C
Drug: Placebo
  Arms: placebo

SUMMARY:
Evaluation of the efficacy of different doses of nor UDCA vs. placebo for the treatment of Primary Sclerosing Cholangitis (PSC). Identification of optimal dose(s)for the treatment of PSC.

DETAILED DESCRIPTION:
Double-blind, randomized, multi-center, placebo-controlled, comparative exploratory phase II-finding trial.The study will be conducted with four treatment groups in the form of a parallel-group comparison and will serve to compare oral treatment with either 500 mg/d, 1000 mg/d or 1500 mg/d norursodeoxycholic acid capsules vs. Placebo capsules for the treatment of PSC.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent
2. Verified diagnosis of PSC
3. PSC patients with or without IBD
4. Women of childbearing potential have to apply during the entire duration of the study a highly effective method of birth control.

Exclusion Criteria:

1. History or presence of other concomitant liver diseases
2. Treatment with UDCA within 8 weeks prior to baseline visit.
3. Child B/C liver cirrhosis
4. Total bilirubin > 3.0 mg/dl at screening or baseline.
5. Any relevant systemic disease
6. TSH>ULN at screening
7. any severe concomitant cardiovascular, renal, endocrine, or psychiatric disorder
8. Any active malignant disease
9. Known intolerance/hypersensitivity to study drug
10. Existing or intended pregnancy of brest feeding
11. Simultaneous participation in another clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2012-12; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in serum AP levels during treatment | 12 weeks

SECONDARY OUTCOMES:
Proportion of patients with at least 50% reduction in s-ALP | 12 weeks

OTHER OUTCOMES:
Adverse Events | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Trauner, Prof, Principal Investigator — Med. Uni Wien; Michael P Manns, Prof, Principal Investigator — Med.Hochschule Hannover
Locations (3):
- Prof. M. Trauner, Vienna, Austria
- Prof. Michael Manns, Hanover, Germany
- Kirsten Boberg, Oslo, Norway

REFERENCES:
- [Derived] Fickert P, Hirschfield GM, Denk G, Marschall HU, Altorjay I, Farkkila M, Schramm C, Spengler U, Chapman R, Bergquist A, Schrumpf E, Nevens F, Trivedi P, Reiter FP, Tornai I, Halilbasic E, Greinwald R, Prols M, Manns MP, Trauner M; European PSC norUDCA Study Group. norUrsodeoxycholic acid improves cholestasis in primary sclerosing cholangitis. J Hepatol. 2017 Sep;67(3):549-558. doi: 10.1016/j.jhep.2017.05.009. Epub 2017 May 18. PMID 28529147